CLINICAL TRIAL: NCT02092012
Title: Comparison of Preemptive Analgesic Effects of Dexketoprofen Versus Dexmedetomidine on the Patients That is Undergoing Abdominal Hysterectomy
Brief Title: Comparison of Preemptive Analgesic Effects of Dexketoprofen Versus Dexmedetomidine on Abdominal Hysterectomy Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, SELDA KAYAALTI, MD, resident, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013/489
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Pain
Keywords: postoperative pain; dexketoprofen trometamol; dexmedetomidine
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — dexketoprofen trometamol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexketoprofen trometamol (Active Comparator): ıv 50 mg dexketoprofen trometamol after anesthesia induction
  Interventions: Drug: dexketoprofen trometamol
- dexmedetomidine (Active Comparator): ıv 1 mcg/kg dexmedetomidine after anaesthesia induction
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: dexketoprofen trometamol — ıv 50 mg dexketoprofen trometamol after anaesthesia induction
  Other Names: arveles
  Arms: dexketoprofen trometamol
Drug: Dexmedetomidine — ıv 1 mcg/kg dexmedetomidine after anaesthesia induction
  Other Names: precedex
  Arms: dexmedetomidine

SUMMARY:
The aim of this study is to investigate comparison of preemptive analgesic effects of dexketoprofen versus dexmedetomidine on the patients that is undergoing abdominal hysterectomy.

DETAILED DESCRIPTION:
Abdominal hysterectomy is associated with moderate to severe postoperative pain which has unfavorable effects on patient's recovery and procedure's outcome. Administration of opioid analgesics is routinely practiced but is limited with dose-related adverse effects.[1] Within this concept, combining an opioid with different analgesics acting by different mechanisms as multimodal analgesia is recommended for effective post-operative pain control Dexketoprofen trometamol is a newly developed, centrally acting NSAID with potency similar to that of μ-opioid agonists.[4] In a number of studies in different pain models, it has been proven to have a good analgesic efficacy and tolerability.

Dexmedetomidine is a highly selective α2 adrenoceptor agonist that provides sedation, analgesia, and sympatholysis. These characteristics make dexmedetomidine useful anesthetic adjunct during operation. Previous studies report that intravenous has a definitive role in postoperative analgesia through the reduction of opioid consumption The aim of this prospective randomized, double-blind study is to evaluate the analgesic efficacy and opioid sparing effects of preemptive single dose of dexketoprofen trometamol in comparison with dexmedetomidine in the patients abdominal hysterectomy , over a 24-hour (h) investigation period.

After institutional approval and informed consent had been obtained, 60 patients scheduled for abdominal hysterectomy randomly allocated into two equal groups. Patients received ıv dexketoprofen 50 mg (Group I), ıv dexmedetomidine 1mcg/kg (Group II) after anesthesia induction and 10 minutes (min) before surgical incision. Patient controlled analgesia was supplied postoperatively using morphine. Hemodynamics, visual analogue scale (VAS), sedation score, morphine consumption, and side effects were recorded every and at 2, 6, 12 and 24 h after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18- 65 year female
* Scheduled for elective abdominal hysterectomy
* No known allergies to drugs
* ASA I-II patients

Exclusion Criteria:

* Pregnancy
* Drug or alcohol abuse
* History of allergic reaction to any of the study drugs
* Ongoing opioid, and non-steroidal anti-inflammatory
* Analgesic therapy
* Cardiac, respiratory, hepatic and/or renal failure
* History of peptic ulcer disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | postoperative 1 day
  Visual Analog Scale on rest and movement record

SECONDARY OUTCOMES:
analgesic consumption | postoperative 1 day
  morphine consumption with patient controlled analgesia record

CONTACTS AND LOCATIONS:
Overall Officials: selda kayaaltı, resident, Principal Investigator — erciyes univercity medicine faculty
Locations (1):
- Erciyes Univercity Medicine Faculty, Kayseri, Turkey (Türkiye)